CLINICAL TRIAL: NCT00824668
Title: A Randomised, Open-labelled, 2-period Crossover Trial Investigating Pharmacodynamics and Pharmacokinetics of Biphasic Insulin Aspart 30 Thrice Daily and Basal-bolus Therapy With Insulin Glargine & Insulin Glulisine in Subjects With Type 2 Diabetes
Brief Title: Comparison of Pharmacodynamics and Pharmacokinetics of Biphasic Insulin Aspart 30 and Insulin Glargine and Insulin Glulisine Therapy in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1832; 2006-006578-92 (EudraCT Number)
Record Dates: First submitted 2009-01-14; First posted 2009-01-19 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Glargine; insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart 30
Drug: insulin glargine
Drug: insulin glulisine

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to compare the 24-hour pharmacodynamics/ pharmacokinetics of biphasic insulin aspart 30 (BiAsp 30) thrice daily treatment with that of a basal-bolus treatment with insulin glargine and insulin glulisine in type 2 diabetic subjects.

Pharmacodynamics is the glucose-lowering effect of the study medication over the entire observation phase from the time of administration and the efficacy period while the pharmacokinetics is the amount of the study insulin that can be determined in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus for 12 months or longer
* Body Mass Index (BMI): 25.0-40.0 kg/m2, both inclusive
* HbA1c between 7.0 and 10.5% at screening
* Insulin treatment for at least 3 months prior to screening with a total daily dose of 0.6 and 0.9 U/kg body weight

Exclusion Criteria:

* Use of any oral antidiabetic agent within the past 2 months
* Cardiac disease: NYHA class III or IV chronic heart failure (CHF), unstable angina, and/or any myocardial infarction (treated or untreated) within 6 months prior to screening
* Hepatic insufficiency (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) equal to or greater than 2 times the central laboratory's upper reference limit)
* Renal insufficiency (serum creatinine equal to or greater than 1.6 mg/dL for males; equal to or greater than 1.4 mg/dL for females)
* Recurrent hypoglycaemia
* Anaemia (haemoglobin less than 13.0 mg/dL in males and less than 12.0 mg/dL in females; WHO-criteria)
* Use of concomitant medications (prescribed or non-prescribed and other than insulin) which may alter glucose metabolism including but not limited to: systemic or inhaled glucocorticoids, anabolic steroids, non-selective beta-blockers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Heise T, Heinemann L, Hovelmann U, Brauns B, Nosek L, Haahr HL, Olsen KJ. Biphasic insulin aspart 30/70: pharmacokinetics and pharmacodynamics compared with once-daily biphasic human insulin and Basal-bolus therapy. Diabetes Care. 2009 Aug;32(8):1431-3. doi: 10.2337/dc09-0097. Epub 2009 Jun 1. PMID 19487640
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com